CLINICAL TRIAL: NCT02428608
Title: A Multi-center, Open Label, Single Dose, Phase II Trial to Demonstrate the Safety of DWP-450 in Adult Subjects for Treatment of Moderate-to-severe Glabellar Lines
Brief Title: Safety Study of DWP-450 (Botulinum Toxin, Type a) to Treat Glabellar Lines - EV-006
Acronym: EV-006
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evolus, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Evolus - CLIN006
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Glabellar Frown Lines
Keywords: Glabellar Lines; Botulinum toxin, Type A
MeSH Terms: interventions — DWP450

STUDY DESIGN:
Masking Description: This is an open label safety study
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botulinum toxin, Tyoe A (Experimental): DWP-450 (Botulinum toxin, Type A)
  Interventions: Biological: DWP-450 (Botulinum purified neurotoxin, Type A)

INTERVENTIONS:
Biological: DWP-450 (Botulinum purified neurotoxin, Type A) — Botulinum toxin, Type A
  Other Names: DWP-450

SUMMARY:
The primary objective is to demonstrate the safety of multiple doses of DWP-450 purified Botulinum neurotoxin, Type A, in treatment of moderate to severe glabellar lines associated with corrugator and procerus muscle activity in adult subjects.

DETAILED DESCRIPTION:
Up to five hundred and thirty (530) subjects will be enrolled and injected with the study drug DWP-450 over the course of the 365 day study.

Subjects with moderate-to-severe glabellar lines at maximum frown on the 4 point Glabellar Line Scale (GLS, 0=none, 1= mild, 2=moderate, 3=severe), as judged by the investigator, will be eligible for injection with DWP-450.

Subjects may receive up to a maximum of 4 treatments and will be followed for 365 days from initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be an adult 18 years of age and over
* Subject is able to provide informed consent and comply with study instructions
* Subject has moderate-to-severe glabellar lines on maximum frown as assessed by the investigator and subject using the GLS
* Subject is willing and able to complete the entire course of the study

Exclusion Criteria:

* Previous treatment with botulinum toxin of any serotype in any area within the last 6 months
* Previous treatment with any facial aesthetic procedure (e.g. injection with fillers, chemical peeling, photo rejuvenation) in the glabellar area within the last 12 months
* Previous insertion of permanent material in the glabellar area
* Planned treatment with botulinum toxin of any serotype in any other body region during the study period
* Any surgery in the glabellar area including surgical removal of the corrugator, procerus, or depressor supercilii muscles or a combination of these, or scars in the glabellar area and the surrounding areas (including eye brow)
* Energy based or cryo-therapy based treatment of facial muscles superior to the lateral canthus
* Any other planned facial aesthetic procedure during the trial period, superior to the level of the lateral canthus (subjects can continue with their usual skin care routine)
* Inability to substantially lessen glabellar frown lines even by physically spreading them apart
* Marked facial asymmetry
* Ptosis of eyelid and/or eyebrow, or history of eyelid and/or eyebrow ptosis
* History of facial nerve palsy
* Excessive dermatochalasis, deep dermal scarring, thick sebaceous skin
* Any active infection in the area of the injection sites
* Medical condition that may affect neuromuscular function (e.g., myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis)
* Evidence of recent alcohol or drug abuse
* Medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study
* Pregnant, nursing or sexually active female subjects who are of childbearing potential and who are not willing to use an acceptable form of contraception
* Known allergy or hypersensitivity to botulinum toxin preparation
* Participation in another interventional clinical study within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rui Avelar, MD, Study Director — Evolus, Inc.
Locations (1):
- The Advanced Skin Research Center at Skin Specialists, PC, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided
Developing a plan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin, Tyoe A
Started | 570
Completed | 487
Not Completed | 83
Not completed — Pregnancy | 2
Not completed — Lost to Follow-up | 37
Not completed — Withdrawal by Subject | 2
Not completed — scheduling conflicts | 15
Not completed — moved away | 10
Not completed — Death | 1
Not completed — various | 16

BASELINE CHARACTERISTICS:
Groups:
- Botulinum Toxin, Type A: DWP-450 (Botulinum toxin, Type A)
  DWP-450 (Botulinum purified neurotoxin, Type A): Botulinum toxin, Type A
Arm/Group | Botulinum Toxin, Type A
Number analyzed (Participants) | 570
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 519
  >=65 years | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 510
  Male | 60

OUTCOME MEASURES:

1. Primary Outcome: The Safety of Repeat DWP-450 Treatments - Proportion of Subjects With at Least One Adverse Event Over 1 Year
Description: The primary safety analysis was the calculation of the proportion of subjects with at least one adverse event that occurred from Day 0 through Day 365.
Time Frame: 365 days
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin, Tyoe A
Number analyzed (Participants) | 570
Participants | 235

2. Other Pre Specified Outcome: Change From Baseline Glabellar Line Scale (GLS) Score at Rest and at Maximum Frown
Description: Proportion of subjects with an improvement of 1 point or more (i.e., ≥1 point responders) on the GLS at rest at end of study/early termination: by Investigator assessment
Time Frame: 365 days
Population: By Investigator assessment, 500 subjects had a GLS score at rest >0 (i.e., 1, 2 or 3) at baseline and therefore could potentially have had a ≥1 point improvement in GLS score at rest at a post-baseline visit; 64 subjects were missing the EOS GLS assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin, Type A
Number analyzed (Participants) | 500
Participants | 355

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Botulinum Toxin, Type A
Serious Adverse Events (participants affected / at risk) | 7/570
Other Adverse Events (participants affected / at risk) | 228/570
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin, Type A (N=570)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin, Type A (N=570)
Headache (Nervous system disorders) | 75 (94)
Migraine (Nervous system disorders) | 4 (6)
Tension headache (Nervous system disorders) | 2 (2)
dizziness (Nervous system disorders) | 1 (1)
hypoaesthesia (Nervous system disorders) | 1 (1)
paraesthesia (Nervous system disorders) | 1 (1)
presyncope (Nervous system disorders) | 1 (1)
radiculitis cervical (Nervous system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 7 (7)
Herpes zoster (Infections and infestations) | 3 (3)
Hordeolum (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 5 (5)
Nasopharyngitis (Infections and infestations) | 13 (16)
Pharyngitis streptococcal (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 14 (15)
Tooth abscess (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 16 (19)
Urinary tract infection (Infections and infestations) | 10 (10)
cellulitis (Infections and infestations) | 1 (1)
conjunctivitis (Infections and infestations) | 1 (1)
cystitis (Infections and infestations) | 1 (1)
diverticulitis (Infections and infestations) | 1 (1)
ear infection (Infections and infestations) | 1 (1)
eye infection (Infections and infestations) | 1 (1)
folliculitis (Infections and infestations) | 1 (1)
gastroenteritis (Infections and infestations) | 1 (1)
genital herpes (Infections and infestations) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
oral herpes (Infections and infestations) | 1 (1)
otitis media (Infections and infestations) | 1 (1)
pharyngitis (Infections and infestations) | 1 (1)
tooth infection (Infections and infestations) | 1 (1)
vaginitis gardnerella (Infections and infestations) | 1 (1)
viral infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 9 (10)
Foot fracture (Injury, poisoning and procedural complications) | 4 (4)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Eye laser scar (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 6 (6)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 6 (6)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Solar lentigo (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1)
Skin swelling (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (2)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1)
mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Blepharospasm (Eye disorders) | 2 (2)
Brow ptosis (Eye disorders) | 3 (3)
Eyelid ptosis (Eye disorders) | 7 (8)
Vision blurred (Eye disorders) | 2 (2)
blepharitis (Eye disorders) | 1 (1)
cataract (Eye disorders) | 1 (1)
chalazion (Eye disorders) | 1 (1)
dry eye (Eye disorders) | 1 (1)
eye swelling (Eye disorders) | 1 (1)
eyelid oedema (Eye disorders) | 1 (1)
eyelid sensory disorder (Eye disorders) | 1 (1)
ocular rosacea (Eye disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 3 (3)
abdominal discomfort (Gastrointestinal disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)
abdominal pain upper (Gastrointestinal disorders) | 1 (1)
diverticulum (Gastrointestinal disorders) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 1 (1)
gastritis (Gastrointestinal disorders) | 1 (1)
large intestine polyp (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
paraesthesia oral (Gastrointestinal disorders) | 1 (1)
salivary gland disorder (Gastrointestinal disorders) | 1 (1)
tooth disorder (Gastrointestinal disorders) | 1 (1)
Injection site bruising (General disorders) | 2 (3)
Injection site pain (General disorders) | 3 (3)
Injection site swelling (General disorders) | 3 (3)
Pyrexia (General disorders) | 3 (5)
fatigue (General disorders) | 1 (1)
injection site pruritus (General disorders) | 1 (1)
injection site reaction (General disorders) | 1 (1)
local swelling (General disorders) | 1 (1)
tenderness (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2)
Bundle branch block right (Cardiac disorders) | 3 (3)
Sinus arrhythmia (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2)
atrioventricular block first degree (Cardiac disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)
supraventricular extrasystoles (Cardiac disorders) | 1 (1)
tachycardia (Cardiac disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 10 (10)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 4 (4)
adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1)
attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Hypersensitivity (Immune system disorders) | 3 (3)
Seasonal allergy (Immune system disorders) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2)
electrocardiogram QT prolonged (Investigations) | 1 (1)
electrocardiogram T wave abnormal (Investigations) | 1 (1)
electrocardiogram abnormal (Investigations) | 1 (1)
intraocular pressure test (Investigations) | 1 (1)
QRS axis abnormal (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2)
hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
breast tenderness (Reproductive system and breast disorders) | 1 (1)
vaginal discharge (Reproductive system and breast disorders) | 1 (1)
vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
hypothyroidism (Endocrine disorders) | 2 (2)
nephrolithiasis (Renal and urinary disorders) | 1 (1)
proteinuria (Renal and urinary disorders) | 1 (1)
menopause (Social circumstances) | 2 (2)
hepatic cyst (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No